CLINICAL TRIAL: NCT05809245
Title: Corneal Neurotization Via Sural Nerve Transfer or Cadaveric Nerve Graft for Neurotrophic Keratopathy
Brief Title: Corneal Neurotization as a Treatment for Neurotrophic Keratopathy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulties with recruitment
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Andrea L Kossler, Director, Oculoplastic Surgery & Orbital Oncology Assistant Professor of Ophthalmology, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 43284
Record Dates: First submitted 2018-05-14; First posted 2023-04-12 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-03

CONDITIONS: Neurotrophic Corneal Ulcer; Neurotrophic Keratitis; Cranial Nerve V Diseases
Keywords: Corneal neurotization; neurotrophic cornea; neurotrophic corneal ulcer
MeSH Terms: conditions — Trigeminal Nerve Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Corneal neurotization (Experimental): Patients will undergo the corneal neurotization as described in the protocol. Their pre and post-procedure corneal sensation will be measured as a primary outcome measure. Secondary outcome measures will include visual acuity, corneal opacity, NEI VFQ, and confocal microscopy.
  Interventions: Procedure: Corneal neurotization

INTERVENTIONS:
Procedure: Corneal neurotization — Autologous sural nerve will be harvested or cadaveric nerve graft will be coapted to an intact sensory branch of the trigeminal nerve. The nerve will be separated into fascicles which will be tunneled under the conjunctiva around the cornea near the limbus.

SUMMARY:
The purpose of this study is to assess the efficacy of sural nerve transfer and cadaveric nerve graft to re-establish corneal sensation in patients with neurotrophic keratopathy.

DETAILED DESCRIPTION:
Corneal anesthesia, which can lead to visually devastating outcomes from ulceration, perforation, and scarring, can be recalcitrant to both medical and surgical treatment[1-3]. Neurotization is a revolutionary technique reported to restore corneal sensation in neurotrophic keratopathy[4-6]. Prior techniques described include direct neurotization with contralateral supraorbital and supratrochlear nerves accessed via a bicoronal incision of the scalp over the forehead[5]; nerve grafting with contralateral supratrochlear nerves accessed via a medial upper eyelid incision[6]; and sural nerve grafting to contralateral supratrochlear nerves accessed via a transverse incision over the medial upper eyelid[4]. Despite the challenges associated with these techniques (needing to subcutaneously tunnel the nerve graft over the nasal bridge or requiring a large bicoronal incision), these techniques all demonstrated efficacy in direct neurotization to improve corneal sensation in these patients.

The investigators aim to assess the efficacy of this innovative surgical technique involving coaptation of the sural nerve or cadaveric nerve allograft to an intact sensory branch of the trigeminal nerve to restore corneal sensation. The investigators have previously described the anatomic feasibility of using the infraorbital nerve using a cadaveric model, of which the results were presented at the American Society of Ophthalmic Plastic and Reconstructive Society Fall meeting in 2017. Utilization of the infraorbital nerve provides advantages over existing techniques due to ease of access via a cosmetically favorable incision, large caliber with increased ability to create a perineural window, relatively short and direct tunnel with possibly more rapid neurotization, and absence of complex surrounding anatomical structures. Others have previously describe success using the contralateral and ipsilateral supraorbital nerve and supratrochlear nerve.

ELIGIBILITY:
Inclusion Criteria:

* Patients with neurotrophic cornea

Exclusion Criteria:

* Patients with history of penetrating keratoplasty

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2018-03-15 (Actual); Primary Completion 2020-02-12 (Actual); Study Completion 2020-02-12 (Actual)

PRIMARY OUTCOMES:
Corneal sensation | Baseline (pre-operative) to 12 months postoperatively
  Corneal sensation will be measured via Cochet Bonnet esthesiometry

SECONDARY OUTCOMES:
Visual acuity | Baseline (pre-operative) to 12 months postoperatively
  Measurement using Snellen eye chart
Corneal opacity | Baseline (pre-operative) to 12 months postoperatively
  Measured based on grade 0-4 based on degree of opacity.

CONTACTS AND LOCATIONS:
Locations (1):
- Andrea Kossler, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ramaesh K, Stokes J, Henry E, Dutton GN, Dhillon B. Congenital corneal anesthesia. Surv Ophthalmol. 2007 Jan-Feb;52(1):50-60. doi: 10.1016/j.survophthal.2006.10.004. PMID 17212990
- [Background] Bonini S, Rama P, Olzi D, Lambiase A. Neurotrophic keratitis. Eye (Lond). 2003 Nov;17(8):989-95. doi: 10.1038/sj.eye.6700616. PMID 14631406
- [Background] Mantelli F, Nardella C, Tiberi E, Sacchetti M, Bruscolini A, Lambiase A. Congenital Corneal Anesthesia and Neurotrophic Keratitis: Diagnosis and Management. Biomed Res Int. 2015;2015:805876. doi: 10.1155/2015/805876. Epub 2015 Sep 16. PMID 26451380
- [Background] Elbaz U, Bains R, Zuker RM, Borschel GH, Ali A. Restoration of corneal sensation with regional nerve transfers and nerve grafts: a new approach to a difficult problem. JAMA Ophthalmol. 2014 Nov;132(11):1289-95. doi: 10.1001/jamaophthalmol.2014.2316. PMID 25010775
- [Background] Terzis JK, Dryer MM, Bodner BI. Corneal neurotization: a novel solution to neurotrophic keratopathy. Plast Reconstr Surg. 2009 Jan;123(1):112-120. doi: 10.1097/PRS.0b013e3181904d3a. PMID 19116544
- [Background] Sepehripour S, Lloyd MS, Nishikawa H, Richard B, Parulekar M. Surrogate Outcome Measures for Corneal Neurotization in Infants and Children. J Craniofac Surg. 2017 Jul;28(5):1167-1170. doi: 10.1097/SCS.0000000000003677. PMID 28570404